CLINICAL TRIAL: NCT05019625
Title: Biomarker Development for Muscular Dystrophies
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Children's Hospital (Other); Wake Forest University (Other); University of Pittsburgh (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Thurman Wheeler, M.D, Physician Scientist, Massachusetts General Hospital
Other Study IDs: 2014P001727
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Myotonic Dystrophy; Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy; Muscular Dystrophy, Duchenne; Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biofluid; muscle tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Single biofluid collection: We will ask eligible volunteers to provide a single urine sample and undergo a single blood draw.
- Serial biofluid and muscle function testing: We will ask eligible volunteers to provide a urine sample, a blood sample, and undergo standard muscle function tests once every six months over a two-year period, and undergo pulmonary function tests and electrocardiogram once per year for two years.
- Biofluid and muscle tissue biopsy: We will ask eligible volunteers to provide a urine sample and undergo a muscle biopsy once.
- Ultrasound and myography testing: We will ask eligible volunteers to provide a single urine sample, a single blood draw, and undergo ultrasound and electrical impedance myography studies once.

SUMMARY:
Current methods of measuring the response to new treatments for muscular dystrophies involve the examination of small pieces of muscle tissue called biopsies. The investigators are interested in finding less invasive methods that reduce the need for muscle biopsies. The purpose of this research is to learn about the possibility of detecting and measuring the activity and severity of muscular dystrophies by examining a urine sample and a blood sample, and some muscles in the arms and legs using tests called ultrasound and electrical impedance myography; both tests are painless and non-invasive. The information that is gathered from this study may help to evaluate, prevent, diagnose, treat, and improve the understanding of human muscle diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with DM1 or DM2 based on genetic testing and/or clinical criteria (some subjects who have positive genetic testing may be asymptomatic, while other subjects who show characteristic clinical features may have declined to have genetic testing done). Control non-DM subjects are unknown to have DM or any other muscular dystrophy by history and may have had no genetic testing.
* Able to provide informed consent or assent for participation in the study.
* Demographic characteristics for single biofluid collection: Males and females age 5 years and older.
* Demographic characteristics for serial biofluid and muscle function testing: Males and females age 14 years and older with DM1.
* Demographic characteristics for biofluid and muscle biopsy: Males and females, ages 18-65 years.

Demographic characteristics for single biofluid collection, ultrasound, and myography: Males and females age 14 years and older.

Exclusion Criteria:

* Medical history of any of the following. State of immunosuppression; coagulopathy; pre-existing liver or kidney disease; documented HIV positive; documented hepatitis B and/or C positive.
* Medications and other drugs. Use of anti-platelet drugs within 7 days prior to blood draw or biopsy; use of anticoagulants within 60 days prior to blood draw or biopsy; active drug or alcohol use or dependence that, in the opinion of the biopsy surgeon, would interfere with post-procedure wound care.
* Other. Inability or unwillingness of the subject to give written informed consent.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Males and females ages 5 years and older with myotonic dystrophy type 1 (DM1), myotonic dystrophy type 2 (DM2), Duchenne muscular dystrophy (DMD), Becker muscular dystrophy (BMD), and facioscapulohumeral muscular dystrophy (FSHD) confirmed by genetic testing or by clinical history and examination are invited to participate. In addition, male and female healthy volunteers ages 18 and older also are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 465 (Estimated)
Dates: Start 2015-02-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Extracellular RNA in biofluids | 6 years
  The extracellular RNA biomarkers in the muscular dystrophy groups will be evaluated and compared with the extracellular RNA content in control groups. Statistical analysis will be used to evaluate the sensitivity and specificity of these markers as measurements of disease activity and severity based on clinical measurements of muscle power, electrocardiogram parameters, pulmonary function test parameters, muscle tissue composition using quantitative ultrasound and electrical impedance myography, and muscle tissue specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Thurman M. Wheeler, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoury L, Hu N, Balaj L, Das S, Georghiou S, Darras B, Clark T, Breakefield XO, Wheeler TM. Analysis of extracellular mRNA in human urine reveals splice variant biomarkers of muscular dystrophies. Nat Commun. 2018 Sep 25;9(1):3906. doi: 10.1038/s41467-018-06206-0. PMID 30254196
- [Background] Antoury L, Hu N, Darras B, Wheeler TM. Urine mRNA to identify a novel pseudoexon causing dystrophinopathy. Ann Clin Transl Neurol. 2019 May 17;6(6):1106-1112. doi: 10.1002/acn3.777. eCollection 2019 Jun. PMID 31211175